CLINICAL TRIAL: NCT03788733
Title: Study of the Efficacy of Melatonin in the Burning Mouth Syndrome
Brief Title: The Efficacy of Melatonin in the Burning Mouth Syndrome
Acronym: BMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Head of Oral Medicine, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University Murcia
Record Dates: First submitted 2018-12-22; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Sleep Disorders, Circadian Rhythm
Keywords: Burning mouth syndrome,; melatonin; pain; sleep
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Burning Mouth Syndrome; Pain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Melatonin ORAL FILM 3mg will be taken by the subject once a day for 8 weeks
  Interventions: Drug: Melatonin 3 mg
- placebo (Placebo Comparator): ORAL FILM 3mg placebo will be taken by the subject once a day for 8 weeks
  Interventions: Drug: Placebo Oral

INTERVENTIONS:
Drug: Melatonin 3 mg — 1 time a day for 8 weeks
  Other Names: melatonin
  Arms: Melatonin
Drug: Placebo Oral — 1 time a day for 8 weeks
  Other Names: Placebo
  Arms: placebo

SUMMARY:
Burning mouth ( BMS) syndrome is the oral disorder characterized by an intraoral burning sensation for which no medical or dental cause can be found. The Headache Classification Committee of the International Headache Society (IHS) defines (BMS) as an ''intraoral burning or dysaesthetic sensation, recurring daily for more than 2 hours per day over more than 3 months, without clinically evident causative lesions''. (BMS) is a common, chronic problem that has a negative impact on quality of life.

A wide variety of medications have been proposed for treating (BMS) both topical and systemic. Unfortunately, no treatment seems to offer assured results. Melatonin is a naturally occurring hormone secreted by the pineal gland. It has soporific effects with oral administration and is well tolerated. It enhances sleep Melatonin also may help sleep disturbances associated with (BMS) ; however, this remains to be proven.

DETAILED DESCRIPTION:
The purpose of this study is to establish whether melatonin can aid in reducing pain improve sleep quality in (BMS)

ELIGIBILITY:
Inclusion Criteria:

* Intraoral burning or dysaesthetic sensation, recurring daily for more than 2 hours per day over more than 3 months, without clinically evident causative lesions

Exclusion Criteria:

* Previous or current therapy with melatonin
* Allergy or hypersensitivity to melatonin
* Less than 18 years old.
* Pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-06-14 (Estimated); Study Completion 2019-12-14 (Estimated)

PRIMARY OUTCOMES:
Sleep Questionnaire | day 0 .The PSQI total score ranges from 0 to 21 with 0 being marvelous sleep and 21 being horrid sleep. The difference score, reported below, is the total score after at least 8 weeks of treatment. A negative score means that the sleep
  The Pittsburgh Sleep Quality Index (PSQI)
Sleep Questionnaire | 8 weeks.The PSQI total score ranges from 0 to 21 with 0 being marvelous sleep and 21 being horrid sleep. The difference score, reported below, is the total score after at least 8 weeks of treatment. A negative score means that the sleep
  The Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
Oral Pain | day 0 .Pain was scored using a Visual Analogue Scale (VAS) (with a score of 1-10: 0 = no pain, 10 = extreme pain)
  Visual Analogue Scale (VAS)
Oral Pain | 8 weeks.Pain was scored using a Visual Analogue Scale (VAS) (with a score of 1-10: 0 = no pain, 10 = extreme pain)
  Visual Analogue Scale (VAS)
Questionnaire ORAL Quality of life | day 0 The instrument consists of 14 items that explore different aspects of oral function and quality of life. The score ranges from 0 to 70, with higher scores corresponding to poorer oral quality of life.
  Questionnaire OHIP 14 Oral quality of life
Questionnaire ORAL Quality of life | 8 weeks The instrument consists of 14 items that explore different aspects of oral function and quality of life. The score ranges from 0 to 70, with higher scores corresponding to poorer oral quality of life.
  Questionnaire OHIP 14 Oral quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Lopez-Jornet Pia, PhD, Principal Investigator — Oral Medicine
Locations (1):
- Lopez-Jornet Pia, Murcia, N/A = Not Applicable, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varoni EM, Lo Faro AF, Lodi G, Carrassi A, Iriti M, Sardella A. Melatonin Treatment in Patients with Burning Mouth Syndrome: A Triple-Blind, Placebo-Controlled, Crossover Randomized Clinical Trial. J Oral Facial Pain Headache. 2018 Spring;32(2):178-188. doi: 10.11607/ofph.1913. PMID 29694465
- [Result] Xie Z, Chen F, Li WA, Geng X, Li C, Meng X, Feng Y, Liu W, Yu F. A review of sleep disorders and melatonin. Neurol Res. 2017 Jun;39(6):559-565. doi: 10.1080/01616412.2017.1315864. Epub 2017 May 1. PMID 28460563